CLINICAL TRIAL: NCT06133387
Title: PARADIGM Study: Prospective Assessment of a Robotic Assisted Device in Gastrointestinal Medicine - En Bloc Trial With the EndoQuest Endoluminal Surgical (ELS) System
Brief Title: PARADIGM - En Bloc Trial With the EndoQuest Endoluminal Surgical (ELS) System
Acronym: PARADIGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EndoQuest Robotics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0001-Rev E
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Lesion; Colorectal Adenoma; Colorectal Polyp; Rectal Lesion; Rectal Adenoma; Rectal Polyp; Sigmoid; Lesion; Sigmoid Colon Polyp
Keywords: Rectal Lesion; Sigmoid Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm 1 (Experimental): * Subjects with benign final pathology and R0 resection is achieved; or,
  * Subjects with benign (but not pre-cancerous) final pathology without R0 resection.
  Subjects in Arm 1 will complete the study after Day 30.
  Interventions: Device: Endoscopic submucosal dissection using the ELS System
- Arm 2 (Experimental): * Subjects with final pathology that is upstaged to cancer; or,
  * Subjects with benign (and pre-cancerous) final pathology without R0 resection.
  Subjects in Arm 2 will undergo 5-year follow-up to assess long-term oncological outcomes including local recurrence, disease-free survival and overall survival.
  Interventions: Device: Endoscopic submucosal dissection using the ELS System

INTERVENTIONS:
Device: Endoscopic submucosal dissection using the ELS System — All subjects will undergo endoscopic submucosal dissection, with or without closure at the discretion of the Investigator, of benign lesions in the rectum and sigmoid colon.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Endoluminal Surgical (ELS) System in subjects undergoing specified transanal endoluminal procedures in the rectum and sigmoid colon. Subjects will undergo endoscopic submucosal dissection (ESD), with or without closure at the discretion of the Investigator, of benign lesions in the rectum and sigmoid colon.

The safety and effectiveness outcomes will be assessed intraoperatively and postoperatively at discharge and Days 7 and 30.

DETAILED DESCRIPTION:
This study will be a prospective, single treatment, multi-center, open-label clinical study. The objective of this study is to evaluate the safety and effectiveness of the ELS System in subjects undergoing specified transanal endoluminal procedures in the rectum and sigmoid colon. Subjects will undergo endoscopic submucosal dissection, with or without closure at the discretion of the Investigator, of benign lesions in the rectum and sigmoid colon (up to 7 cm in size and up to 75% of the colorectal circumference).

The safety and effectiveness outcomes will be assessed intraoperatively and postoperatively at discharge, Day 7 (-2 +7 days) and Day 30 (-7 +14 days).

Subjects with lesions resected using the study device will be allocated into two different study arms:

Arm 1:

* Subjects with benign final pathology and R0 resection is achieved; or,
* Subjects with benign (but not pre-cancerous) final pathology without R0 resection.

Arm 2:

* Subjects with final pathology that is upstaged to cancer; or,
* Subjects with benign (and pre-cancerous) final pathology without R0 resection.

Subjects in Arm 1 will complete the study after Day 30. Arm 1 subjects in which R0 resection was not achieved should receive routine care, including any additional treatment as needed at the discretion of the physician, even if occurring after study exit at Day 30. Any non-study-related care of Arm 1 subjects occurring after study exit may be performed by the Investigator or transferred to another physician at the discretion of the Investigator and will not be collected for this trial.

Subjects in Arm 2 will undergo 5-year follow-up to assess long-term oncological outcomes including local recurrence, disease-free survival and overall survival.

To ensure a total of 50 subjects are included in the final analysis, the study may enroll up to 56 subjects at up to 5 clinical sites in the U.S. No individual site will be permitted to enroll more than 60% of the subjects in the final data set to ensure that a single site does not dominate the results and analysis. Enrollment will end when 50 subjects have completed 30-day follow-up or the maximum enrollment number has been reached, whichever occurs first.

In addition to the total number of enrolled subjects, each Investigator will enroll up to 2 lead-in cases. Lead-in cases will be analyzed separately in the final clinical study report.

ELIGIBILITY:
Preoperative Inclusion Criteria:

1. Subject is ≥22 years at the time of consent.
2. Subject has a BMI ≤ 50 kg/m2.
3. Subject has an ASA score of ≤ 3.
4. Subject has benign lesion(s) of the rectum or sigmoid colon, such as adenoma (with low- or high-grade dysplasia), neuroendocrine tumor, or other type of polyp as assessed by the most recent colonoscopy/flexible sigmoidoscopy.
5. Subject has lesion ≤ 7 cm in size (dimension of greatest extent) and ≤ 75% of the colorectal circumference as assessed by the most recent colonoscopy/flexible sigmoidoscopy.
6. Subject is eligible for standard endoscopic submucosal dissection.
7. Subject agrees to participate in the study by giving signed informed consent.

Preoperative Exclusion Criteria:

1. Subject anatomy is unsuitable for endoscopic visualization or endoluminal surgery.
2. Subject has a history of inflammatory bowel disease.
3. Subject has an untreated active infection at the time of the procedure.
4. Subject is considered part of a vulnerable population (e.g., prisoners, mentally disabled).
5. Subject has a severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions (e.g., cancer).
6. Subject is breastfeeding or pregnant or intends to become pregnant during the study.
7. Subject is currently enrolled in or discontinued within the last 30 days from a clinical trial of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
8. Subject with EF ≤ 45, high cardiac or high pulmonary risk (these subjects require clearance from a cardiologist and pulmonologist, as applicable).
9. Subject on preoperative blood thinners, such as coumadin or heparin, that cannot be weaned prior to surgery.
10. Subject is moderately or severely immunocompromised.
11. In the opinion of the Investigator, the subject is unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.

Intraoperative Exclusion Criteria (assessed with third-party endoscope):

1. Inadequate bowel prep.
2. Complex anatomical findings not feasible for an endoluminal approach.
3. Anatomical narrowing distal to the lesion site.
4. Lesion not located in the rectum or sigmoid colon.
5. Lesion size >7 cm (dimension of greatest extent) or occupies >75% of the colorectal circumference.
6. Lesion demonstrates characteristics indicative of invasive carcinoma, such as failure to lift upon submucosal injection, or any other features that raise the Investigator's suspicion of cancer.

   Intraoperative Exclusion Criteria (assessed with study device):
7. In the opinion of the Investigator, the subject and/or subject anatomy is not suitable for study device use for any reason.
8. Lesion location not accessible by the study device.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
En Bloc Resection Rate | On Day 0 (day of procedure)
  The percentage of target lesions across all subjects that are excised in a single specimen.
ESD-Related Complication-Free Rate | From enrollment to Day 30.
  The percentage of subjects free from study device-related bleeding and perforation complications intraoperatively and postoperatively through Day 30.

SECONDARY OUTCOMES:
R0 Resection Rate | On Day 0 (day of procedure)
  The percentage of target lesions across all subjects that are resected with lateral and deep margins free of residual disease under microscopic visualization.
Conversion-Free Rate | On Day 0 (day of procedure)
  The percentage of intended resections that do not require conversion to achieve successful completion of the resection.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - AdventHealth, Orlando, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - HCA Healthcare, Houston, Texas